CLINICAL TRIAL: NCT05319600
Title: Does a Behavior Change Skills and Physical Activity Program Improve Self-regulation and Health Outcomes in Adolescents With Type 1 Diabetes?
Brief Title: Technology-delivered Physical Activity Program for Adolescents With Type 1 Diabetes
Acronym: Activate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Amy Hughes Lansing, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001482; P20GM103644 (NIH)
Record Dates: First submitted 2022-03-25; First posted 2022-04-08 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes
Keywords: adolescents; physical activity intervention; diabetes self-management; behavior-change skills training
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Adolescents (aged 13-17) diagnosed with type 1 diabetes will all complete a baseline assessment where they will be randomized to complete a 12-week physical activity and behavior-change skills training intervention, or to follow their usual diabetes care plan for 12 weeks. Both groups will receive a Garmin fitness activity tracker wrist watch to track their physical activity over the 12-week study period. Follow-up assessments for all participants will take place after 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm will complete an intervention delivered remotely via an online website and online communication from the research team across the 12-week intervention period. This intervention has two parts, taking place simultaneously over the 12 weeks. First, participants will complete 8 web-delivered online behavior-change skills learning sessions which include reading and activities. Second, participants will be given daily and weekly personalized physical activity goals to meet, which will be tracked via their Garmin activity tracker and weekday text and if indicated video support. They have the opportunity to win money each week for meeting activity goals.
  Interventions: Behavioral: Diabetes behavior change skills training; Behavioral: Physical activity promotion program
- Treatment as usual - Control (No Intervention): This arm will not complete an intervention. Participants will be instructed to wear a Garmin activity tracker but will be given no other specific instructions, other than to continue to follow their normal daily diabetes care plan.

INTERVENTIONS:
Behavioral: Diabetes behavior change skills training — Behavior-change skills training will be provided through eight web-delivered content and activity sessions across the 12-week program. Sessions 1 through 4 will occur weekly and sessions 5 through 8 biweekly. Each session takes approximately 15-20 minutes for the adolescent to complete both content learning and related activities. These learning sessions focus on skills like problem solving and goal setting.
  Arms: Intervention
Behavioral: Physical activity promotion program — The physical activity incentives program includes 12 weeks of personalized goals and incentives for increasing physically active minutes along with weekday text-based support. Active minutes, defined as minutes with moderate to vigorous physical activity, will be tracked via a Garmin fitness activity tracker.
  Arms: Intervention

SUMMARY:
This project is comprised of a two-arm randomized control trial (RCT) testing the feasibility, acceptability, and preliminary efficacy of a nationally scalable program, Activate, a 12-week, technology-delivered diabetes behavior-change skills training and physical activity promotion program for adolescents with type 1 diabetes. The researchers have a recruitment goal of 30 participants, but will enroll beyond 30 to address any withdrawal and ensure sample size is met. A primary goal of the study is assessing the feasibility and acceptability of the program, which combines two previously piloted components. Then, the investigators will compare the 12-week Activate program to a treatment as usual control group on proximal outcomes of behavior-change skills and daily active minutes. The investigators will also explore the impact of the Activate program on secondary mechanisms and outcomes linked with later type 1 diabetes health disparities: adolescent diabetes behavior regulation, psychological distress, inflammation, glycemic outcomes, and cardiovascular disease risk. It is hypothesized that a diabetes behavior-change skills training and physical activity intervention will be acceptable, and effective at improving behavior-change skills and daily active minutes, as well as other mechanisms and outcomes linked with later type 1 diabetes health disparities.

DETAILED DESCRIPTION:
Adolescents with type 1 diabetes and socioeconomic disadvantage experience significant health disparities in glycemic outcomes in adolescence and cardiovascular disease and diabetes-related death later in adulthood. Socioeconomic disadvantage is associated with elevated glycosylated hemoglobin (HbA1c) and 3x risk of repeat hospitalizations for diabetic ketoacidosis as well as 2-3x risk of cardiovascular disease and diabetes-related death. Suboptimal glycemic outcomes are a powerful determinant of long-term health complications and costs, with a 1% reduction in HbA1c contributing to up to a 40% reduction in risk for later nephropathy, retinopathy, and macrovascular disease. Given the substantial health disparities for persons with type 1 diabetes and socioeconomic disadvantage and the many challenges that adolescents face with achieving optimal glycemic levels (<20% nationally meet American Diabetes Association HbA1c targets), this is a critical population to support in health behavior change via psychosocial intervention during adolescence. Unfortunately, existing evidence-based psychosocial type 1 diabetes interventions for adolescents, including robust multi-system approaches, have demonstrated limited efficacy for behavior change that results in improved glycemic outcomes and none have directly targeted cardiovascular health outside of glycemic outcomes. In this project, the researchers pursue a new avenue for intervention innovation by testing a nationally-scalable diabetes behavior-change skills training and physical activity intervention program to improve glycemic outcomes and decrease cardiovascular disease risks for adolescents with type 1 diabetes including those with socioeconomic disadvantage .

In this study the researchers will conduct a two-arm randomized trial with 30 adolescents with type 1 diabetes, comparing the 12-week Activate program to a treatment-as-usual control group. This study has 2 primary aims. First, the investigators will assess acceptability of the Activate program by examining participant engagement with the Activate program components. To assess the preliminary efficacy of the Activate program the investigators will examine changes in proximal outcomes of behavior-change skills (goal setting, problem-solving, and coping skills), and active minutes compared between treatment and control groups from baseline to a 12-week follow-up assessment. Second, the investigators will explore the impact of the Activate program on secondary mechanisms and outcomes linked with longer-term type 1 diabetes health disparities.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13-17 years old
* At least 18 months post-diagnosis for type 1 diabetes
* Parent reported moderate to no physical activity for adolescent
* Ability to complete measures and intervention program in English
* Access to broadband or cellular internet
* Resides in and receives healthcare in the United States

Exclusion Criteria:

* Ward of state
* Active psychosis
* Severe medical or psychiatric illness that limit participation (including any contraindications for physical activity)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Hughes Lansing, PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No
Overall analyses and de-identified data can be shared as described in participant consent, however, individual participant data will not be shared.

REFERENCES:
- [Background] Wood JR, Miller KM, Maahs DM, Beck RW, DiMeglio LA, Libman IM, Quinn M, Tamborlane WV, Woerner SE; T1D Exchange Clinic Network. Most youth with type 1 diabetes in the T1D Exchange Clinic Registry do not meet American Diabetes Association or International Society for Pediatric and Adolescent Diabetes clinical guidelines. Diabetes Care. 2013 Jul;36(7):2035-7. doi: 10.2337/dc12-1959. Epub 2013 Jan 22. PMID 23340893
- [Background] Clements MA, Foster NC, Maahs DM, Schatz DA, Olson BA, Tsalikian E, Lee JM, Burt-Solorzano CM, Tamborlane WV, Chen V, Miller KM, Beck RW; T1D Exchange Clinic Network. Hemoglobin A1c (HbA1c) changes over time among adolescent and young adult participants in the T1D exchange clinic registry. Pediatr Diabetes. 2016 Aug;17(5):327-36. doi: 10.1111/pedi.12295. Epub 2015 Jul 8. PMID 26153338
- [Background] Menzin J, Korn JR, Cohen J, Lobo F, Zhang B, Friedman M, Neumann PJ. Relationship between glycemic control and diabetes-related hospital costs in patients with type 1 or type 2 diabetes mellitus. J Manag Care Pharm. 2010 May;16(4):264-75. doi: 10.18553/jmcp.2010.16.4.264. PMID 20433217
- [Background] Effect of intensive diabetes treatment on the development and progression of long-term complications in adolescents with insulin-dependent diabetes mellitus: Diabetes Control and Complications Trial. Diabetes Control and Complications Trial Research Group. J Pediatr. 1994 Aug;125(2):177-88. doi: 10.1016/s0022-3476(94)70190-3. PMID 8040759
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Hood KK, Rohan JM, Peterson CM, Drotar D. Interventions with adherence-promoting components in pediatric type 1 diabetes: meta-analysis of their impact on glycemic control. Diabetes Care. 2010 Jul;33(7):1658-64. doi: 10.2337/dc09-2268. PMID 20587726
- [Background] Ellis DA, Templin T, Naar-King S, Frey MA, Cunningham PB, Podolski CL, Cakan N. Multisystemic therapy for adolescents with poorly controlled type I diabetes: Stability of treatment effects in a randomized controlled trial. J Consult Clin Psychol. 2007 Feb;75(1):168-74. doi: 10.1037/0022-006X.75.1.168. PMID 17295576
- [Background] Stanger C, Lansing AH, Scherer E, Budney A, Christiano AS, Casella SJ. A Web-Delivered Multicomponent Intervention for Adolescents with Poorly Controlled Type 1 Diabetes: A Pilot Randomized Controlled Trial. Ann Behav Med. 2018 Nov 12;52(12):1010-1022. doi: 10.1093/abm/kay005. PMID 30418521
- [Derived] Cashmore BA, Cooper TE, Evangelidis NM, Green SC, Lopez-Vargas P, Tunnicliffe DJ. Education programmes for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD007374. doi: 10.1002/14651858.CD007374.pub3. PMID 39171639

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric endocrinology clinic and type 1diabetes community advertisements nationally.
Period: Overall Study
Arm/Group | Intervention | Treatment as Usual - Control
Started | 17 | 14
Completed | 16 | 10
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Population: 1 subject who withdrew from the study was excluded from analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Treatment as Usual - Control | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.31 (1.25) | 15.00 (1.41) | 14.63 (1.35)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 8 | 6 | 14
  Transgender | 2 | 1 | 3
  Do not identify as female, male, or transgender | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 9 | 6 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 1 | 1
  Hispanic/Latino | 1 | 0 | 1
  White | 14 | 13 | 27
  Two or more races | 1 | 0 | 1
Length since diagnosis [Mean (Standard Deviation); unit: years] | 5.33 (2.68) | 6.92 (2.42) | 6.07 (2.65)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Physical Activity
Description: The Garmin fitness activity tracker tracking will be used to determine the average number of daily minutes with moderate to vigorous physical activity, metabolic equivalents (METs) greater than or equal to 3 METs.
Time Frame: daily for all days from week 1 through week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Intervention | Treatment as Usual - Control
Number analyzed (Participants) | 16 | 14
minutes | 209.08 [105.49 to 312.66] | 79.84 [-30.91 to 190.59]
Statistical Analysis 1: Comparison: Intervention vs Treatment as Usual - Control; Test type: Superiority — treatment group as predictor baseline-residualized week 12 scores in linear regression; p < 0.05, Regression, Linear; Slope = 129.2, 95% CI 2-sided [-22.52 to 280.98], Standard Error of Mean 73.96 — Control coded as 0 and treatment as 1

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Intervention | Treatment as Usual - Control
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 0/17 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT05319600/Prot_001.pdf
  • Statistical Analysis Plan (2024-12-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT05319600/SAP_002.pdf
  • Informed Consent Form (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT05319600/ICF_000.pdf